CLINICAL TRIAL: NCT03887702
Title: A Phase III Randomized Trial of Prophylactic Antiviral Therapy in Patients With Current or Past Hepatitis B Virus (HBV) Infection Receiving Anti-Cancer Therapy for Solid Tumors
Brief Title: Prophylactic Antiviral Therapy in Patients With Current or Past Hepatitis B Virus Infection Receiving Anti-Cancer Therapy for Solid Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to accrue
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S1614; NCI-2018-00592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1614 (Other: SWOG); SWOG-S1614 (Other: DCP); S1614 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis B Infection; Malignant Solid Neoplasm
MeSH Terms: conditions — Hepatitis B | interventions — Practice Guidelines as Topic; Standard of Care; entecavir; tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (TAF, TDF, entecavir: prophylactic) (Experimental): [Cohort 1] Patients receive TAF PO QD or TDF PO QD or entecavir PO QD immediately or within 42 days after initial dose of chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entecavir; Drug: Tenofovir Alafenamide; Drug: Tenofovir Disoproxil Fumarate
- Arm 2 (TAF, TDF, entecavir: upon indication) (Experimental): [Cohort 1] Patients receive TAF PO QD or TDF PO QD or entecavir PO QD after HBV reactivation during chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entecavir; Drug: Tenofovir Alafenamide; Drug: Tenofovir Disoproxil Fumarate
- Arm 3 (TAF, TDF, entecavir: upon indication) (Experimental): [Cohort 2] Patients receive TAF PO QD or TDF PO QD or entecavir PO QD after HBV reactivation during chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entecavir; Drug: Tenofovir Alafenamide; Drug: Tenofovir Disoproxil Fumarate
- Arm 4 (Anti-Viral therapy: usual care) (Active Comparator): [Cohort 2] Patients receive anti-HBV therapy at the discretion of the physician. Any Food and Drug Administration (FDA) approved anti-viral medication for treatment of HBV may be utilized.
  Interventions: Other: Best Practice; Drug: Entecavir; Drug: Tenofovir Alafenamide; Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Other: Best Practice — Receive best practice
  Other Names: standard of care; standard therapy
  Arms: Arm 4 (Anti-Viral therapy: usual care)
Drug: Entecavir — Given PO
  Other Names: Baraclude; BMS-200475-01; ETV; SQ-34676; SQ34676
Drug: Tenofovir Alafenamide — Given PO
  Other Names: GS 7340; GS-7340; TFV Alafenamide
Drug: Tenofovir Disoproxil Fumarate — Given PO
  Other Names: PMPA Prodrug; TDF; Tenofovir DF; Viread

SUMMARY:
This phase III trial studies the effect of hepatitis B antiviral (anti-HBV) therapy in preventing liver complications in patients with chronic or past hepatitis B virus (HBV) who are receiving anti-cancer therapy for solid tumors. People with chronic or past HBV who are undergoing therapy for cancer are at an increased risk for changes in the liver which could be minor or severe. Anti-HBV therapy acts against infections caused by HBV and may help reduce the chance that HBV gets worse or comes back in patients receiving anti-cancer therapy for solid tumors.

DETAILED DESCRIPTION:
Co-Primary Objectives

1. To compare the effect of prophylactic anti-HBV therapy versus upon indication anti-HBV therapy on time-to-adverse liver outcomes of liver failure or liver-related death in patients with chronic HBV infection (HBsAg+ and anti-HBc+) receiving anti-cancer therapy for solid tumors.
2. To compare the effect of upon indication anti-HBV therapy versus usual care on time-to-adverse liver outcomes of liver failure or liver-related death in patients with past HBV infection (HBsAg- and anti-HBc+) receiving anti-cancer therapy for solid tumors.

Secondary Objectives

1. Using time-to-event analysis, to compare the effect of anti-HBV therapy versus upon indication anti-HBV therapy on HBV reactivation, on the combined endpoint of adverse liver outcomes (liver failure or liver-related death) and HBV reactivation, and on HBV flare by arm in patients with chronic HBV infection receiving anticancer therapy for solid tumors.
2. Using time-to-event analysis, to compare the effect of upon indication anti-HBV therapy versus usual care on HBV reactivation, on the combined endpoint of adverse liver outcomes (liver failure or liver-related death) and HBV reactivation, and on HBV flare by arm in patients with past HBV infection receiving anti-cancer therapy for solid tumors.

Translational Objectives

1. To compare baseline and changes in overall immune status and HBV-specific immune response in patients with solid tumors and chronic or past HBV infection receiving anti-cancer therapy, and to compare the differences in these immune responses by HBV reactivation status.
2. To identify demographic and clinical predictors and correlative immunologic biomarkers of HBV reactivation after receipt of anti-cancer therapy in patients with solid tumors and chronic or past HBV infection.

OUTLINE: Patients are recruited in two cohorts (Cohort 1: chronic HBV infection, Cohort 2: past HBV infection), with each cohort randomized equally to one of two potential treatment arms.

Chronic HBV Infection (Cohort 1) Arms:

Arm 1: Patients receive tenofovir alafenamide (TAF) orally (PO) once daily (QD) or tenofovir disoproxil fumarate (TDF) PO QD or entecavir PO QD immediately or within 42 days after initial dose of chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.

Arm 2: Patients receive TAF PO QD or TDF PO QD or entecavir PO QD after HBV reactivation during chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.

Past HBV infection (Cohort 2) Arms:

Arm 3: Patients receive TAF PO QD or TDF PO QD or entecavir PO QD after HBV reactivation during chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.

Arm 4: Patients receive anti-HBV therapy at the discretion of the physician. Any Food and Drug Administration (FDA) approved anti-viral medication for HBV may be used.

(Cohort 1: Arm 2 and Cohort 2: Arm 3 follow the same treatment plan, but are considered part of separate parallel studies and are therefore identified as separate arms.)

Patients are followed for 24 months: every 4 weeks from randomization to week 24, then every 8 weeks thereafter up to week 104.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with stage I-III solid tumor malignancy; patients with only carcinoma in situ or with stage IV disease are excluded
* Patients must not have lymphoma, leukemia, or myeloma
* Patients must not have primary liver cancer, known cirrhosis, or evidence of any malignancy that involves the liver
* Patients must be planning to receive systemic anti-cancer therapy (either single agent or some combination of systemic cytotoxic therapy, systemic immunotherapy or systemic targeted therapy) for this solid tumor
* Patients must not have been previously treated with the same anti-cancer therapy regimen that is now anticipated; the anti-cancer therapy does not have to be first-line therapy; prior and/or concurrent radiotherapy is allowed
* Patients must be registered <= 28 days prior to the planned start date of anti-cancer therapy; if the patient has started systemic anti-cancer therapy, patient must be registered <= 42 days after the initiation of first cycle of anti-cancer therapy
* Patients who have received prior anti-cancer therapy must have discontinued all previous therapies (excluding planned anti-cancer therapy to occur in conjunction with this study) >= 1 day prior to registration to this study
* Patients must not have had any cancer therapy regimen that includes anti-CD20
* Patients must not be receiving antiviral medications active against HBV, including: adefovir, entecavir, lamivudine, telbivudine, tenofovir disoproxil fumarate, tenofovir alafenamide (TAF), or any other Food and Drug Administration (FDA) approved agents for the treatment of hepatitis B; patients who have previously received antiviral medication must not have required any antiviral medication active against HBV >= 90 days prior to registration to this study
* Patients must not have had hematopoietic stem cell transplantation therapy
* Patients must not be taking or planning to take warfarin
* Patients who will be treated with TAF must not be taking or planning to take oxcarbazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine, or St. John's Wort
* Patients who will be treated with TAF and are concomitantly taking or plan to take carbamazepine must be given an increased dose of TAF or alternatively be given ETV or TDF
* Patients must have results for the following HBV tests done within 28 days prior to registration: HBsAg AND anti-HBc (total immunoglobulin [Ig] or IgG, but not IgM only) AND hepatitis B surface antibody (anti-HBs); for the anti-HBs test, quantitative or qualitative (including "indeterminate") results are allowable
* Patients must have tested positive for HBsAg or anti-HBc (total Ig, IgG, but not IgM) and must have baseline HBV deoxyribonucleic acid (DNA) completed <= 42 days prior to registration
* Complete blood count (CBC) must be completed <= 28 days prior to registration; results do not need to be in the institutional limits of normal
* International normalized ratio (INR) must be completed <= 28 days prior to registration; results must <= 1.2 x institutional limits of normal
* Alanine aminotransferase (ALT) must be obtained <= 28 days prior to registration; ALT must be < 1.5 x institutional ULN
* Total bilirubin must be obtained <= 28 days prior to registration; total bilirubin must be < 1.5 x institutional ULN
* Creatinine results must be obtained <= 28 days prior to registration
* Patients must not have known current active hepatitis C infection (HCV); active HCV is defined by a detectable HCV ribonucleic acid (RNA) level; Note: HCV testing is not required for eligibility
* Patients must not have a history of human immunodeficiency (HIV) infection; patients with unknown HIV status must have HIV testing completed <= 365 days prior to registration
* Patients must have Zubrod performance status of 0-2
* Patients must not be pregnant or nursing, as the safety of the study drug in pregnant and nursing women has not been established; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must have specimens collected for submission as outlined
* Patients must be offered the opportunity to participate in optional translational medicine studies as outlined
* Patients with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)
* Patients may have concurrent participation in other clinical trials that entail cytotoxic, immunotherapy, targeted therapy; surgical treatment; radiotherapy treatment; or any combination thereof
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P Hwang, Principal Investigator — SWOG Cancer Research Network
Locations (193):
- United States (192):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Broward Health North, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - Kaiser Permanente Washington, Seattle, Washington
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 4 (Anti-Viral Therapy: Usual Care): [Cohort 2] Patients receive anti-HBV therapy at the discretion of the physician. Any Food and Drug Administration (FDA) approved anti-viral medication for HBV may be used.
Period: Overall Study
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
Started (This represents the number of participants registered to the arms.) | 0 | 0 | 2 | 2
Received Anti-HBV Treatment Per Assignment (This represents the number of participants who actually received any anti-viral HBV therapy on their assigned study arm (Arms 2 and 3 are upon indication; Arm 4 is physician discretion with any anti-HBV therapy allowed)) | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 2
Not completed — Study terminated | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: There were no participants registered to the Chronic HBV infection cohort [Cohort 1, Arms 1 and 2]
Groups:
- Arm 1 (TAF, TDF, Entecavir: Prophylactic): [Cohort 1] Patients receive tenofovir alafenamide (TAF) orally (PO) once daily (QD) or tenofovir disoproxil fumarate (TDF) PO QD or entecavir PO QD immediately or within 42 days after initial dose of chemotherapy. Treatment continues for up to 6 months after the last dose of chemotherapy or a maximum of 24 months in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care) | Total
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] |  |  | 47.5 [45.5 to 49.5] | 75.4 [64.4 to 86.3] | 62.45 [45.5 to 86.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 2 | 1 | 3
  Male |  |  | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 0 | 0 | 0
  Not Hispanic or Latino |  |  | 2 | 2 | 4
  Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0 | 0
  Asian |  |  | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 1 | 1
  Black or African American |  |  | 0 | 0 | 0
  White |  |  | 0 | 0 | 0
  More than one race |  |  | 0 | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Liver Outcome
Description: Adverse liver outcome: Defined as liver-related death or liver failure (ascites, hepatic encephalopathy or impaired hepatic synthetic function defined as total bilirubin ≥ 5 mg/dL or INR ≥ 2.0) not due to disease progression in the liver. Assessment of the primary endpoint will be made by sites and subsequently adjudicated by the research oversight team by blinded review.
Time Frame: From randomization to 24 months
Population: There were no participants registered to the Chronic HBV infection cohort [Cohort 1, Arms 1 and 2]
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
Number analyzed (Participants) | 0 | 0 | 2 | 2
Participants |  |  | 0 | 0

2. Secondary Outcome: Number of Participants With Hepatitis B Virus (HBV) Reactivation
Description: HBV reactivation is is defined as one of the following:
  * ≥ 2 log (100-fold) increase in HBV DNA compared to baseline in patients with detectable HBV DNA at baseline, or
  * HBV DNA ≥ 3 log (1,000) IU/mL in a patient with previously undetectable HBV DNA, or
  * HBV DNA ≥ 4 log (10,000) IU/mL if baseline HBV DNA not available, or
  * HBsAg seroreversion (HBsAg- to HBsAg+) in a patient previously HBsAg-.
Time Frame: From randomization up to 24 months
Population: There were no participants registered to the Chronic HBV infection cohort [Cohort 1, Arms 1 and 2]
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
Number analyzed (Participants) | 0 | 0 | 2 | 2
Participants |  |  | 0 | 0

3. Secondary Outcome: Number of Participants With Hepatitis B Virus (HBV) Flare
Description: Hepatitis flare is defined as ALT > 3 x baseline and >100 U/L.
Time Frame: From randomization to 24 months
Population: There were no participants registered to the Chronic HBV infection cohort [Cohort 1, Arms 1 and 2]
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
Number analyzed (Participants) | 0 | 0 | 2 | 2
Participants |  |  | 0 | 0

4. Secondary Outcome: Combined Endpoint of Adverse Liver Outcomes and HBV Reactivation, Number of Participants
Description: Adverse liver outcome: Defined as liver-related death or liver failure (ascites, hepatic encephalopathy or impaired hepatic synthetic function defined as total bilirubin ≥ 5 mg/dL or INR ≥ 2.0) not due to disease progression in the liver. Assessment of the primary endpoint will be made by sites and subsequently adjudicated by the research oversight team by blinded review.
  HBV reactivation is defined as one of the following:
  * ≥ 2 log (100-fold) increase in HBV DNA compared to baseline in patients with detectable HBV DNA at baseline, or
  * HBV DNA ≥ 3 log (1,000) IU/mL in a patient with previously undetectable HBV DNA, or
  * HBV DNA ≥ 4 log (10,000) IU/mL if baseline HBV DNA not available, or
  * HBsAg seroreversion (HBsAg- to HBsAg+) in a patient previously HBsAg-.
  The combined endpoint of adverse liver outcomes and HBV reactivation is the occurrence of either adverse liver outcome or HBV reactivation as defined above.
Time Frame: From randomization to 24 months
Population: There were no participants registered to the Chronic HBV infection cohort [Cohort 1, Arms 1 and 2]
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
Number analyzed (Participants) | 0 | 0 | 2 | 2
Participants |  |  | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 2 years, but, with the exception of study endpoints, adverse events were only collected after participants began treatment with anti-HBV therapy.
Description: No participants received experimental treatment on this study. No participants were registered in the Chronic HBV cohort [Cohort 1]. In the Past HBV cohort [Cohort 2]:
  * no participants assigned to Arm 3 experienced HBV reactivation, which would have prompted treatment with the study-assigned anti-HBV therapy according to protocol
  * one participant in Arm 4 (standard of care) began anti-HBV therapy at physician discretion.
Arm/Group | Arm 1 (TAF, TDF, Entecavir: Prophylactic) | Arm 2 (TAF, TDF, Entecavir: Upon Indication) | Arm 3 (TAF, TDF, Entecavir: Upon Indication) | Arm 4 (Anti-Viral Therapy: Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
On November 15, 2022, the study was discontinued with no further follow-up required after it was determined that the accrual goal could not be met. Four participants had been accrued to Cohort 2 and no participants to Cohort 1. No adverse liver events, hepatitis B flares, or hepatitis B reactivations had occurred at the time the study was discontinued. As a result, planned time-to-event analyses for these outcomes could not be completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03887702/Prot_SAP_000.pdf